CLINICAL TRIAL: NCT04962217
Title: Experiences Among Family Members, Carers and Significant Others of Brief Admission by Self-referral for Self-harming and Suicidal Persons: a Qualitative Study
Brief Title: Experiences of Brief Admission From the Perspective of Family and Significant Others
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Sofie Westling, associate professor, Region Skane
Other Study IDs: 2019-02557
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Suicidal Ideation; Self Injurious Behavior Without Suicidal Intent; Self-Harm, Deliberate
MeSH Terms: conditions — Suicidal Ideation; Self-Injurious Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Semi-structured interviews — Each participant will attend a 30-60 minute semi-structured interview conducted by the CI

SUMMARY:
As a result of a randomized controlled trial (NCT02985047) BA is continuously offered to persons with self-harm at risk for suicide in Skåne, Sweden. This qualitative inductive study aims to provide experiences among family members, carers and significant others of Brief Admission by self-referral for self-harming and suicidal persons based on individual semi-structured interviews. Participants will be identified through suggestion from persons with an active BA contract. Interviews, estimated to last 30-60 minutes, will be analyzed by a phenomenological hermeneutic method or by content analysis depending on richness and depth in the interviews. Findings from this study will be published.

DETAILED DESCRIPTION:
As a result of the randomized controlled trial evaluating BA in Skåne (NCT02985047), BA is since January 2019, continuously offered to persons with self-harm at risk for suicide in Skåne, Sweden. Parallel to the clinical trial qualitative interview studies have been performed on the experiences of BA, with participants during the pilot phase of the trial and among the most severely ill persons and from the viewpoint of psychiatric staff. The present study aims to complement the above-mentioned studies with analysis of real-life experiences of BA from the perspective of loved ones to persons with current access to BA. This is important since the persons close to those suffering from recurrent self-harm and suicidal ideation play an essential role in times of crisis and may beneficially contribute to motivation as well as effects of provided care.

In this qualitative inductive study individual semi-structured interviews will be held with family members, carers and significant others of persons with an active BA contract, who has given informed consent to participate. To identify potential informants, persons with an active BA contract, who have used BA within the last three months, at the wards in Lund, Malmö, Helsingborg or Kristianstad will be contacted and asked about contact information (name and telephone number) to a person close to them who may be contacted regarding inclusion in the present study. A variation of contract length (minimum one month since first signed contract) is strived for. The number of interviews will depend on the number of active contracts at the included wards and the proportion of those where potential participants may be contacted and who subsequently consent to participate, but with a maximum of 25 interviews. Interviews are estimated to be 30-60 minutes, and will be conducted in a calm place, chosen by the participant. Interviews will be performed by doctoral students in psychiatry and supervised by a senior researcher with experience of psychiatry and qualitative research. Interviews will be transcribed and analyzed by a phenomenological hermeneutic method or by content analysis depending on richness and depth in the interviews. Findings from this study will be published.

ELIGIBILITY:
Inclusion Criteria:

* Family member, carer or significant other as defined by persons with access to Brief Admission by self-referral through one of the psychiatric departments in Skåne, Sweden (Lund, Malmö, Helsingborg or Kristianstad).
* At least 18 years of age.
* Able to consent to study participation through written and oral information.
* Given consent to participate

Exclusion Criteria:

* below the age of 18.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Family member, carer or significant other as defined by persons with access to Brief Admission by self-referral through one of the psychiatric departments in Skåne, Sweden (Lund, Malmö, Helsingborg or Kristianstad).
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Lived experiences | 60 minutes
  Data from semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Westling, PhD, Principal Investigator — Region Skåne
Locations (1):
- Psykiatri och habilitering, Region Skåne, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have no ethical approval to share data from interviews.